CLINICAL TRIAL: NCT03934112
Title: Impact of Transfusional Practice on the Morbidity and Mortality of Patients in Intensive Care
Brief Title: Impact of Transfusional Practice on the Morbidity and Mortality of Patients in Intensive Care Unit
Acronym: PATMORE
Status: Recruiting | Type: Observational
Sponsor: Centre Hospitalier Universitaire de Besancon (Other)
Responsible Party: Sponsor
Other Study IDs: API/2016/72
Record Dates: First submitted 2019-04-26; First posted 2019-05-01 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Transfusion Related Complication

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This study will allow correlating transfusion monitoring and patients' prognostic according to the chosen outcome criteria.

These data could thus represent a basis for transfusion recommendations, except for intensive care and vital emergencies.

It will also bring information about the actual transfusion monitoring in intensive care unit (ICU), in the period following the stay in the ICU and after hospital discharge.

ELIGIBILITY:
Inclusion criteria:

* Patient admitted to medical and surgical resuscitation units of Besançon and Dijon university hospitals, all causes considered
* Patient admitted between 1st January 2012 to 31st December 2017

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All patients treated in medical and surgical resuscitation units of Besançon and Dijon university hospitals during the study period (from 01/01/2012 to 31/12/2017) are concerned.
Sampling Method: Probability Sample
Enrollment: 150000 (Estimated)
Dates: Start 2020-01-03 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Survival at 90 days after leaving ICU | Day 90
  All-cause mortality 90 days after leaving ICU

CONTACTS AND LOCATIONS:
Locations (1):
- CHU de Besançon, Besançon, France